CLINICAL TRIAL: NCT02486302
Title: A PROSPECTIVE, MULTICENTER NON-INTERVENTIONAL STUDY TO EVALUATE THE EFFICACY OF ENBREL (REGISTERED) (ETANERCEPT) OVER A PERIOD OF 12 MONTHS IN THE ROUTINE TREATMENT OF PATIENTS WITH RHEUMATOID ARTHRITIS, AXIAL SPONDYLOARTHRITIS, PSORIATIC ARTHRITIS, OR PLAQUE PSORIASIS WITH PARTICULAR FOCUS ON THE CLINICAL STATUS IMPROVEMENTS STILL OBSERVABLE AFTER 12 WEEKS OF TREATMENT
Brief Title: A Study To Evaluate The Efficacy Of Enbrel (REGISTERED) Etanercept Over A Period Of 12 Months In The Routine Treatment Of Patients With Rheumatoid Arthritis, Axial Spondyloarthritis, Psoriatic Arthritis, Or Plaque Psoriasis.
Acronym: ADEQUATE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801385; ADEQUATE (Other: Alias Study Number)
Record Dates: First submitted 2015-06-28; First posted 2015-07-01 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Axial Spondyloarthritis; Plaque Psoriasis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Axial Spondyloarthritis | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation Group
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept shall be used according to clinical practice and in line with the summary of product characteristics.

SUMMARY:
The purpose of this non-interventional study is to evaluate the efficacy of etanercept during routine clinical use over a maximum of 12 months in patients with rheumatoid arthritis (RA), psoriatic arthritis(PsA), axial spondyloarthritis(axSpA) or plaque psoriasis (PsO). In so doing, particular attention will be paid to the proportion of those patients who only attain the desired treatment goal after 12 weeks of treatment. The primary efficacy end point for the study is the proportion of patients who attain the desired treatment goal after 12 and 24 weeks,

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of RA, axSpA, PsA or PsO
* No prior treatment with etanercept and eligibility for treatment with etanercept according to the summary of product characteristics.

Exclusion Criteria:

* The contraindications, special warnings, and precautions according to the summary of product characteristics for etanercept shall apply.
* The additional documentation of the patient in another post-marketing study with etanercept is not permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory and Hospital care patients treated for Rheumatoid Arthritis, Axial Spondyloarthritis, Psoriasis Arthritis or Plaque Psoriasis in Germany
Sampling Method: Non-Probability Sample
Enrollment: 1534 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (180):
- Germany (180):
  - Rheumatologisches MVZ Dresden GmbH im Gesundheitszentrum Dresden - Klotzsche (GZDK), Dresden, Saxony
  - private practise Hemmerich, Aachen
  - private practise Kurthen, Aachen
  - Gesundheits- und Pflegezentrum Alsfeld gGmbH, Alsfeld
  - private practise Kupka, Altenburg
  - Private Practise Boehm, Altenholz
  - Private Practise Marycz, Amberg
  - Klinikum Bad Bramstedt, Bad Bramstedt
  - private practise Gause, Bad Bramstedt
  - private practise Messis, Bad Homburg
  - ACURA Rheumazentrum Bad Kreuznach, Bad Kreuznach
  - private practise Hesse, Bad Kreuznach
  - private practise Manger, Bamberg
  - private practise Balzer, Bautzen
  - private practise Winkler, Bautzen
  - private practise Ochs, Bayreuth
  - private practise Schmitt-Haendle, Bayreuth
  - Charité Berlin Rheumatologie und Klinische Immunologie, Berlin
  - Med. Versorgungszentrum Ambulantes Gesundheitszentrum Charite Campus Mitte, Berlin
  - private practise Hasert, Berlin
  - Praxis Roßbacher, Berlin
  - private practise Bozorg, Berlin
  - private practise Brandt-Jürgens, Berlin
  - private practise Herzberg, Berlin
  - private practise Remstedt, Berlin
  - private practise Seifert, Berlin
  - private practise Zinke, Berlin
  - private practise Kors, Berlin
  - Rheumaklinik Berlin-Buch, Berlin
  - private practise Miehe, Berlin
  - private practise Schnorfeil, Berlin
  - private practise Koelnberger, Bogen
  - private practise Barth, Borna
  - private practise Eisterhues, Braunschweig
  - Private Practise Ramaker-Brunke, Braunschweig
  - private practise Mall, Bremen
  - private practise Schwichtenberg, Bremen
  - Private Practise Wagener, Bruchhausen-Vilsen
  - private practise Feuchtenberger, Burghausen
  - private practise Budde, Bückeburg
  - Mvz Agliomed, Chemnitz
  - private practise Schneider, Chemnitz
  - private practise Wilden, Cologne
  - Office of Parysa Alborz, MD, Cologne
  - private practise Geißler, Cottbus
  - private practise Kirrstetter, Deggendorf
  - Kreiskrankenhaus Demmin GmbH, Demmin
  - private practise Heidlas, Dessau
  - private practise Bebnowski, Dortmund
  - private practise Gerlach, Dresden
  - private practise Lüthke, Dresden
  - private practise Fischer, Dresden
  - private practise Oppers, Dresden
  - private practise Roch, Dresden
  - private practise Fendler, Duisburg
  - private practise Riesopp, Duisburg
  - private practise Strothmeyer, Düsseldorf
  - Bezirksklinikum Obermain, Ebensfeld
  - private practise Berendt, Eberswalde
  - private practise Pech, Eberswalde
  - Asklepios MVZ Nord SH GmbH, c/o AK St. Georg, Elmshorn
  - Elbe Elster MVZ GmbH, Elsterwerda
  - MVZ Kaestner + Kaestner GbR, Erfurt
  - private practise Koch, Erfurt
  - Universitaetsklinikum Essen, Klinik fuer Dermatologie, Essen
  - private practise Freitag, Falkensee
  - private practise Häckel, Frankenberg
  - private practise Fritzsch, Frankfurt
  - Klinikum der J.W. Goethe-Universität, Klinik für Dermatologie, Klinische Forschung, Frankfurt am Main
  - private practise Höhne, Fraureuth
  - private practise Müller, Freiberg
  - private practise Behringer, Fulda
  - private practise Bussmann, Geilenkirchen
  - private practise Zeh, Geislingen A.d. Steige
  - Private Practice Abahji, Germering
  - Private Practise, Giessen
  - Praxis Dres. Dr.Brinkmann, Schult, Samimi-Fard, Gladbeck
  - private practise Schumann, Groß Reken
  - private practise Kühne, Haldensleben I
  - private practise Liebhaber, Halle
  - MVZ Rheumatologie und Autoimmunmedizin GmbH, Hamburg
  - MVZ Nord GmbH, Hamburg
  - Katholisches Marienkrankenhaus Geriatrische Klinik, Hamburg
  - Private Practise Höhle, Hamburg
  - private practise Dahmen, Hamburg
  - private practise Weinhardt, Hamburg
  - private practise Aries, Hamburg
  - Praxis Praxis Dr. Szabo & Kollegen, Hamm
  - Private Practise Stille, Hanover
  - private practise Stein, Hanover
  - private practise Heilig, Heidelberg
  - private practise Lassak-Siedl, Heidelberg
  - Universitätsklinikum Heidelberg, Heidelberg
  - private Practise Pawlak, Heilbad Heiligenstadt
  - private practise Schleußner, Heilbad Heiligenstadt
  - private practise Thies, Herrsching am Ammersee
  - private practise Meier, Hofheim
  - private practise Wernicke, Hohen Neuendorf
  - Private Practice Streibl, Holzkirchen
  - private practise Kapelle, Hoyerswerda
  - Uniklinik Jena, Jena
  - Private Practise Kremers, Jülich
  - private practise Bräunig, Kahla
  - Praxis Mauer, Kamenz
  - Private Practise Turin, Karlstadt am Main
  - private practise Schwab, Kiel
  - private practise Merkel, Königs Wusterhausen
  - private practise Straub, Kronach
  - Kreiskrankenhaus Langenau, Langenau
  - Boche-Hamann-Teich, Leipzig
  - private practise Schwarze, Leipzig
  - private practise Zeiger, Leipzig
  - private practise Wiemers, Leipzig
  - private practise Weiß, Lichtenstein
  - private practise Holst, Ludwigslust
  - Private Practise Legler, Lübeck
  - private practise Kudela, Magdeburg
  - private practise Raschke, Magdeburg
  - private practise Sieburg, Magdeburg
  - private practise Weimann, Magdeburg
  - Hautklinik der Universitätsmedizin Mainz KöR,Clinical Research Center, Mainz
  - private practise Zimmermann, Malchow
  - Praxis Roßbach, Mansfeld OT Großörner
  - private practise Harmuth, Marktredwitz
  - Private Practise Bödekker, Marl
  - private practise Reck, Mittelherwigsdorf
  - private practise Vollmer, Mönchengladbach
  - private practise Krüger, München
  - Stadt Klinikum Muenchen, München
  - private practise Raub, Münster
  - private practise Berger, Naunhof
  - private practise Klopsch, Neubrandenburg
  - Rheumazentrum SH Mitte GbR, Neumünster
  - private practise Scholz, Neustadt-Glewe
  - private practise Kloos, Neuwied
  - Private Practise Hein, Nienburg
  - Private Practise Vogel, Nuremberg
  - private practise Albert, Offenburg
  - private practise Voglau, Oldenburg
  - private practise Gräßler, Pirna
  - private practise Welcker, Planegg
  - private practise Baumann, Plauen
  - Private Practise Petersen, Potsdam
  - Rheumahaus Potsdam GbR, Potsdam
  - Knappschaftskrankenhaus Püttlingen, Püttlingen
  - private practise Wassenberg, Ratingen
  - private practise Schwokowski, Ratzeburg
  - private practise Rumpel, Regensburg
  - Private Practise Walter, Rendburg
  - Private Practise Kotterik, Reutlingen
  - Private Practise Hoene, Rostock
  - private practise Richter, Rostock
  - private practise Lankow, Rostock
  - private practise Biewer, Saarbrücken
  - Private Practise Mobius, Schwerin
  - private practise Möbius, Schwerin
  - private practise Ständer, Schwerin
  - private practise Melzer, Seesen
  - Company for Medical Study&Service Selters, Selters/Ww
  - Private Practise Hoese, Stadthagen
  - private practise Steinborn, Straubing
  - private practise Engel, Stuttgart
  - ZIRS - Zentrum für Interdisziplinäre Rheumatologie Stuttgart, Stuttgart
  - Private Practice Fahr, Suhl
  - private practise Pyra, Torgelow
  - MVZ der Johanniter, Treuenbrietzen
  - Praxis Dr. Haas, Tübingen
  - Private Practice Jacki, Tübingen
  - Universitätsklinikum Tübingen, Tübingen
  - Berufsausübungsgemeinschaft Dr. med Petra Roll und Dr. Margarete Kratzsch, Ulm / Donau
  - private practise Rinaldi, Ulm / Donau
  - Praxis Dres. Winkler-Gyulay, Moeller, Unna
  - private practise Otte, Wesel
  - private practise Schuart, Wissen/ Luhe
  - private practise Metz, Wittstock
  - private practise Senger, Wunstorf
  - Klinikverbund St. Antonius und St. Josef GmbH, Krankenhaus St. Josef, Wuppertal
  - Private Practise Sprekeler, Zeven
  - private practise Fricke-Wagner, Zwickau
  - private practise Alliger, Zwiesel

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Feist E, Baraliakos X, Behrens F, Thaci D, Plenske A, Klaus P, Meng T. Etanercept in Axial Spondyloarthritis, Psoriatic Arthritis, and Plaque Psoriasis: Real-World Outcome Data from German Non-interventional Study ADEQUATE. Rheumatol Ther. 2024 Apr;11(2):331-348. doi: 10.1007/s40744-023-00633-2. Epub 2024 Feb 3. PMID 38308727
- [Derived] Feist E, Baraliakos X, Behrens F, Thaci D, Klopsch T, Plenske A, Blindzellner LK, Klaus P, Meng T, Loschmann PA. Effectiveness of Etanercept in Rheumatoid Arthritis: Real-World Data from the German Non-interventional Study ADEQUATE with Focus on Treat-to-Target and Patient-Reported Outcomes. Rheumatol Ther. 2022 Apr;9(2):621-635. doi: 10.1007/s40744-021-00418-5. Epub 2022 Feb 3. PMID 35113363
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801385&StudyName=A%20Prospective%2C%20Multicenter%20Non-interventional%20Study%20To%20Evaluate%20The%20Efficacy%20Of%20Enbrel%20%28registered%29%20%28etanercept%29%20Over%20A%20Period%20Of%2012%20Months%20In%20The%20Routine%20Treatment%20Of%20Patients%20With%20Rheumatoid%20Arthritis%2C%20Axial%20Spondyloarthritis%2C%20Psoriatic%20Arthritis%2C%20Or%20Plaque%20Psoriasis%20With%20Particular%20Focus%20On%20The%20Clinical%20Status%20Improvements%20Still%20Observable%20After%2012%20Weeks%20Of%20Treatment

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: All participants with rheumatoid arthritis (RA), axial spondyloarthritis (axSpA), psoriatic arthritis (PsA), or plaque psoriasis (PsO) taking etanercept in the routine treatment as per clinical practice and in line with summary of product characteristics clinical, were observed for a period of 12 months.
Period: Overall Study
Arm/Group | Etanercept
Started | 1534
Treated | 1523
Completed | 858
Not Completed | 676
Not completed — Discontinued prematurely | 410
Not completed — Documentation not completed | 255
Not completed — Excluded due to legal reasons | 8
Not completed — Not treated | 3

BASELINE CHARACTERISTICS:
Population: Treated set included all documented participants who were treated, had at least 1 post-baseline value and had an adverse event (AE) documented.
Groups:
- Etanercept: All participants with RA, axSpA, PsA, or PsO taking etanercept in the routine treatment as per clinical practice and in line with summary of product characteristics clinical, were observed for a period of 12 months.
Arm/Group | Etanercept
Number analyzed (Participants) | 1465
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There is no information available for age for 6 participants (=missing values).
  years
    number analyzed (Participants) | 1459
    (all) | 54.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 901
  Male | 564
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Rheumatoid Arthritis (RA) Who Achieved 28 Joint Disease Activity Score (DAS28) Less Than (<) 2.6 at Week 12
Description: Disease activity score based on 28-joints count (DAS28) calculated as weighted average of swollen joint count (SJC) and tender joint count (TJC) using the 28 joints count, erythrocyte sedimentation rate (ESR) (millimeter per hour [mm/h]) and patient's global assessment (PtGA) of disease activity (recorded on a visual analog scale [VAS] scale of 0 mm-100 mm, where 0 = no disease activity and 100=high disease activity). DAS28 <2.6 = remission, DAS28 less than or equal to (<=) 3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Week 12
Population: Per-protocol (PP) set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with RA evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Etanercept: All participants with RA taking etanercept in the routine treatment as per clinical practice and in line with summary of product characteristics clinical, were observed for a period of 12 months.
Arm/Group | Etanercept
Number analyzed (Participants) | 794
Participants | 194

2. Primary Outcome: Number of Participants With Rheumatoid Arthritis (RA) Who Achieved 28 Joint Disease Activity Score (DAS28) Less Than (<) 2.6 at Week 24
Description: DAS28 calculated as weighted average of SJC and TJC using the 28 joints count, ESR [mm/h] and PtGA of disease activity (recorded on a VAS scale of 0 mm-100 mm, where 0 = no disease activity and 100=high disease activity). DAS28<2.6 = remission, DAS28 <=3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Week 24
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with RA evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 664
Participants | 203

3. Primary Outcome: Number of Participants With Rheumatoid Arthritis (RA) Who Achieved 28 Joint Disease Activity Score (DAS28) Less Than (<) 2.6 at Week 12 and Maintained Till 52 Weeks
Description: as for outcome 2
Time Frame: Week 12 up to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 147
Participants | 58

4. Primary Outcome: Number of Participants With Rheumatoid Arthritis (RA) Who Achieved 28 Joint Disease Activity Score (DAS28) Less Than (<) 2.6 at Week 24 and Maintained Till 52 Weeks
Description: as for outcome 2
Time Frame: Week 24 up to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 169
Participants | 88

5. Primary Outcome: Number of Participants With PsO Who Achieved 75% Improvement From Baseline in Psoriasis Area & Severity Index(PASI75) Score or Physician's Global Assessment(PGA) of Clear or Almost Clear And Dermatology Life Quality Index(DLQI) Total Score of 0 or 1
Description: PASI:combined assessment of lesion severity & area affected into single score as: 0(no disease)-72(maximal disease). Body divided into=head,upper/lower limbs,trunk;each area scored & scores combined for final PASI. For each section % area of skin involved was estimated:0(0%)-6(90-100%) & severity estimated by clinical signs of erythema,induration,desquamation; range 0(none)-4(very marked). Final PASI=sum of severity parameters for each section*area score*weighing factor(head=0.1,upper limbs=0.2,trunk=0.3,lower limbs=0.4). PASI75:>=75% reduction in PASI from Baseline. PGA psoriasis:average assessment of erythema,induration,desquamation of all psoriatic lesions, scored on 5-point scale: 0(no psoriasis)-4(severe disease). Clear & almost clear indicate score 0 or 1. DLQI:10-item questionnaire, measures impact of skin disease on participant's quality of life. Each question evaluated on 4-point scale as: 0(not at all)-3 (very much). Total DLQI score:0(no effect)-30(extremely large effect).
Time Frame: Week 12
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with PsO.
Measure: Count of Participants; unit: Participants
Groups:
- Etanercept: All participants with PsO taking etanercept in the routine treatment as per clinical practice and in line with summary of product characteristics clinical, were observed for a period of 12 months.
Arm/Group | Etanercept
Number analyzed (Participants) | 70
Participants | 5

6. Primary Outcome: Number of Participants With Axial Spondyloarthritis (axSpA) Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) Less Than (<) 1.3 at Week 12
Description: ASDAS is a score combining the assessment of back pain, peripheral pain/swelling, duration of morning stiffness, PtGA (all assessed on a VAS (0-100cm, where 0 = no disease activity and 100=high disease activity), CRP (mg/L). ASDAS ranged as inactive disease: 0 <= ASDAS < 1.3; moderate disease activity: 1.3 <= ASDAS < 2.1; high disease activity: 2.1 <= ASDAS <= 3.5; very high disease activity: 3.5 < ASDAS.
Time Frame: Week 12
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with axSpA evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Etanercept: All participants with axSpA taking etanercept in the routine treatment as per clinical practice and in line with summary of product characteristics clinical, were observed for a period of 12 months.
Arm/Group | Etanercept
Number analyzed (Participants) | 200
Participants | 38

7. Primary Outcome: Number of Participants With Psoriatic Arthritis (PsA) Who Achieved Either 28 Joint Disease Activity Score (DAS28) Less Than (<) 2.6 or Met Minimal Disease Activity (MDA) Criteria at Week 12
Description: DAS28 calculated as average of from SJC and TJC using the 28 joints count, ESR (mm/h), PtGA of disease activity (recorded on a VAS scale of 0 mm-100 mm, where 0 = no disease activity and 100=high disease activity). DAS28<2.6 = remission, DAS28 <=3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity. A participant was classified as MAD if the participant met at least 5 of 7 following criteria: 1) TJC <=1; 2) SJC =<1; 3) PASI <= 1 or body surface area (BSA) <=3; 4) Participant pain on VAS <= 15 (assessed pain using a 0 mm - 100 mm VAS scale where 0 mm = minimum possible pain [best] and 100 mm = maximum possible pain [worst]; 5) PtGA on VAS <= 20 (all assessed on a VAS 0-100cm, where 0 = no disease activity and 100=high disease activity); 6) Health assessment questionnaire disability index (HAQ-DI) <= 0.5(HAQ=3.16-[0.028* hannover functional questionnaire [FFbH]); 7) Tender enthesial points <= 1.
Time Frame: Week 12
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with PsA evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Etanercept: All participants with PsA taking etanercept in the routine treatment as per clinical practice and in line with summary of product characteristics clinical, were observed for a period of 12 months.
Arm/Group | Etanercept
Number analyzed (Participants) | 240
Participants | 92

8. Primary Outcome: Number of Participants With Plaque Psoriasis (PsO) Who Achieved 75% Improvement in Psoriasis Area and Severity Index (PASI75) Score or a Physician's Global Assessment (PGA) of "Clear" or "Almost Clear" and DLQI Total Score of 0 or 1 at Week 24
Description: as for outcome 5
Time Frame: Week 24
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with PsO evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 59
Participants | 11

9. Primary Outcome: Number of Participants With Axial Spondyloarthritis (axSpA) Achieving Ankylosing Spondylitis Disease Activity Score (ASDAS) Less Than (<) 1.3 at Week 24
Description: as for outcome 6
Time Frame: Week 24
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 152
Participants | 28

10. Primary Outcome: Number of Participants With Psoriatic Arthritis (PsA) Achieving Either 28 Joint Disease Activity Score (DAS28) Less Than (<) 2.6 or Met Minimal Disease Activity (MDA) Criteria at Week 24
Description: DAS28 calculated as average of SJC and TJC using the 28 joints count, ESR (mm/h) and PtGA of disease activity (recorded on a VAS scale of 0 mm-100 mm, where 0 = no disease activity and 100=high disease activity). DAS28<2.6 = remission, DAS28 <=3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity. A participant was classified as MAD if the participant met at least 5 of 7 following criteria: 1) TJC t<=1; 2) SJC =<1; 3) PASI <= 1 or BSA <=3; 4) Participant pain on VAS <= 15 (assessed pain using a 0 mm - 100 mm VAS scale where 0 mm = minimum possible pain [best] and 100 mm = maximum possible pain [worst]; 5) PtGA on VAS <= 20 (all assessed on a VAS 0-100cm, where 0 = no disease activity and 100=high disease activity); 6) HAQ-DI <= 0.5(HAQ=3.16-[0.028*FFbH); 7) Tender enthesial points <= 1.
Time Frame: Week 24
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 209
Participants | 106

11. Secondary Outcome: Percentage of Participants Who Continued With Treatment up to Weeks 12, 24, 36 and 52: Treated Set (TS)
Time Frame: Baseline up to Weeks 12, 24, 36, 52
Population: Treated set included all documented participants who were treated, had at least 1 post-baseline value and had an AE documented.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1465
percentage of participants
  Up to Week 12 | 89.5
  Up to Week 24 | 81.2
  Up to Week 36 | 75.6
  Up to Week 52 | 71.6

12. Secondary Outcome: Percentage of Participants Who Continued With Treatment up to Weeks 12, 24, 36 and 52: Per-Protocol (PP) Set
Time Frame: Baseline up to Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1453
percentage of participants
  Up to Week 12 | 89.4
  Up to Week 24 | 81.1
  Up to Week 36 | 75.6
  Up to Week 52 | 71.6

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) up to Weeks 12, 24, 36 and 52: Treated Set
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were measured up to Week 12, 24, 36 and 52 of exposure with study drug that were absent before treatment or that worsened relative to pretreatment state. TEAEs included both SAEs and non-SAEs.
Time Frame: Baseline up to Weeks 12, 24, 36, 52
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1465
Participants
  Up to Week 12 | 417
  Up to Week 24 | 567
  Up to Week 36 | 651
  Up to Week 52 | 699

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events up to Weeks 12, 24, 36 and 52: Per-Protocol (PP) Set
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were measured up to Week 12, 24, 36 and 52 of exposure with study drug that were absent before treatment or that worsened relative to pretreatment state. TEAEs included both SAEs and non-SAEs.
Time Frame: Baseline up to Weeks 12, 24, 36, 52
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1453
Participants
  Up to Week 12 | 416
  Up to Week 24 | 564
  Up to Week 36 | 646
  Up to Week 52 | 694

15. Secondary Outcome: Number of Participants Achieving 28 Joint Disease Activity Score (DAS28) Remission at Weeks 12, 24, 36 and 52
Description: DAS28 calculated as average of from SJC and TJC using the 28 joints count, ESR (mm/h), PtGA of disease activity (recorded on a VAS scale of 0 mm-100 mm, where 0 = no disease activity and 100=high disease activity). DAS28<2.6 = remission, DAS28 <=3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity. Participants who had DAS28 <= 2.6 were considered in remission.
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with RA or PsA. "Number analyzed" signifies participants analyzed for this outcome measure at specified time points.
Measure: Count of Participants; unit: Participants
Groups:
- Etanercept: All participants with RA or PsA taking etanercept in the routine treatment as per clinical practice and in line with summary of product characteristics clinical, were observed for a period of 12 months.
Arm/Group | Etanercept
Number analyzed (Participants) | 1078
Participants
  Week 12: number analyzed (Participants) | 1034
  Week 12 | 278
  Week 24: number analyzed (Participants) | 873
  Week 24 | 305
  Week 36: number analyzed (Participants) | 742
  Week 36 | 263
  Week 52: number analyzed (Participants) | 663
  Week 52 | 271

16. Secondary Outcome: Patient Global Assessment of Disease Activity (PtGA) Scores at Weeks 12, 24, 36 and 52
Description: Participants answered question: "How do you assess your current disease activity?" Participants responded by using a 0 - 100 mm visual analog scale where 0 mm = no activity and 100 mm = highest possible activity.
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. "Number analyzed" signifies participants analyzed for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 1453
mm
  Week 12: number analyzed (Participants) | 1224
  Week 12 | 39.8 (24.9)
  Week 24: number analyzed (Participants) | 1048
  Week 24 | 35.5 (25.1)
  Week 36: number analyzed (Participants) | 906
  Week 36 | 32.7 (23.8)
  Week 52: number analyzed (Participants) | 791
  Week 52 | 30.5 (23.3)

17. Secondary Outcome: Mean Visual Analogue Scale (VAS) Fatigue Scores at Weeks 12, 24, 36 and 52
Description: Participants assessed their fatigue using a 0 - 100 mm VAS, where 0 mm = no fatigue and 100 mm = worst possible fatigue.
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 1453
mm
  Week 12: number analyzed (Participants) | 1245
  Week 12 | 40.9 (30.1)
  Week 24: number analyzed (Participants) | 1036
  Week 24 | 37.7 (29.5)
  Week 36: number analyzed (Participants) | 902
  Week 36 | 36.1 (28.9)
  Week 52: number analyzed (Participants) | 789
  Week 52 | 33.5 (27.8)

18. Secondary Outcome: Mean Visual Analogue Scale (VAS) Pain Scores at Weeks 12, 24, 36 and 52
Description: Participants assessed pain using a 0 mm - 100 mm VAS scale where 0 mm = minimum possible pain (best) and 100 mm = maximum possible pain (worst).
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Number analyzed signifies participants analyzed for this outcome at specified time points.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 1453
mm
  Week 12: number analyzed (Participants) | 1236
  Week 12 | 38.3 (26.9)
  Week 24: number analyzed (Participants) | 1045
  Week 24 | 34.9 (26.3)
  Week 36: number analyzed (Participants) | 901
  Week 36 | 32.9 (25.6)
  Week 52: number analyzed (Participants) | 791
  Week 52 | 31.1 (24.7)

19. Secondary Outcome: Physician Global Assessment (PGA) of Disease Activity Scores at Weeks 12, 24, 36 and 52
Description: PGA of Disease Activity was measured on a 0 to 100 mm VAS, with 0 mm = no disease activity; 100 mm= high disease activity.
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 1453
mm
  Week 12: number analyzed (Participants) | 1365
  Week 12 | 32.5 (21.1)
  Week 24: number analyzed (Participants) | 1137
  Week 24 | 26.9 (20.5)
  Week 36: number analyzed (Participants) | 990
  Week 36 | 23.8 (19.4)
  Week 52: number analyzed (Participants) | 891
  Week 52 | 21.7 (18.9)

20. Secondary Outcome: Patient Health Quessionare-2 (PHQ-2) Scores at Weeks 12, 24, 36 and 52
Description: The PHQ-2 is a brief depression screening instrument and enquire two factors: frequency of depressed mood and anhedonia (inability to feel pleasure in normally pleasurable activities) over the past 2 weeks, scoring each question on scale of 0 ("not at all") to 3 ("nearly every day"). Total PHQ-2 score ranged from 0-6 (0 indicate not at all: depression/anhedonia can be ruled out; 6 indicate nearly every day: worsening of depression/anhedonia).
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1453
units on a scale
  Week 12: number analyzed (Participants) | 1315
  Week 12 | 2.0 (1.6)
  Week 24: number analyzed (Participants) | 1102
  Week 24 | 1.8 (1.6)
  Week 36: number analyzed (Participants) | 952
  Week 36 | 1.7 (1.5)
  Week 52: number analyzed (Participants) | 830
  Week 52 | 1.6 (1.5)

21. Secondary Outcome: Rheumatoid Arthritis(RA): Spearman Correlation Coefficient Between Patient Global Assessment (PtGA) of Disease Activity, VAS Fatigue, VAS Pain Score, Patient Health Quessionare-2 (PHQ-2) and PGA of Disease Activity at Weeks 12, 24, 36, 52
Description: The PtGA of disease activity was measured on a VAS ranged from 0 mm to 100 mm, where 0 = no disease activity and 100=high disease activity. Participants assessed their fatigue during the last 7 days using a 0 mm - 100 mm VAS, where 0 mm = no fatigue and 100 mm = worst possible fatigue. Participants assessed pain using a 0 mm - 100 mm VAS where 0 mm = minimum possible pain (best) and 100 mm = maximum possible pain (worst). The PHQ-2 is a brief depression screening instrument and enquire two factors: frequency of depressed mood and anhedonia over the past 2 weeks, scoring each question on scale of 0 ("not at all") to 3 ("nearly every day"). Total PHQ-2 ranged from 0-6. PGA disease activity was measured on a 0 mm to 100 mm VAS, with 0 mm = no disease activity and 100mm = maximum possible disease activity. Correlation coefficient between each of these parameters was measured using spearman correlation coefficient and reported.
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with RA. "Number analyzed" signifies participants analyzed for this outcome measure at specified time points.
Measure: Number (95% Confidence Interval); unit: spearman correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 824
spearman correlation coefficient
  Week 12: PtGA versus (vs.) Fatigue: number analyzed (Participants) | 684
  Week 12: PtGA versus (vs.) Fatigue | 0.514 [0.456 to 0.567]
  Week 12: PtGA vs. Pain: number analyzed (Participants) | 686
  Week 12: PtGA vs. Pain | 0.825 [0.799 to 0.847]
  Week 12: PtGA vs. PHQ-2: number analyzed (Participants) | 681
  Week 12: PtGA vs. PHQ-2 | 0.450 [0.387 to 0.507]
  Week 12: PtGA vs. PGA: number analyzed (Participants) | 670
  Week 12: PtGA vs. PGA | 0.603 [0.552 to 0.649]
  Week 12: Fatigue vs. Pain: number analyzed (Participants) | 689
  Week 12: Fatigue vs. Pain | 0.586 [0.535 to 0.633]
  Week 12: Fatigue vs. PHQ-2: number analyzed (Participants) | 693
  Week 12: Fatigue vs. PHQ-2 | 0.577 [0.525 to 0.624]
  Week 12: Fatigue vs. PGA: number analyzed (Participants) | 683
  Week 12: Fatigue vs. PGA | 0.370 [0.303 to 0.433]
  Week 12: Pain vs. PHQ-2: number analyzed (Participants) | 686
  Week 12: Pain vs. PHQ-2 | 0.529 [0.473 to 0.581]
  Week 12: Pain vs. PGA: number analyzed (Participants) | 676
  Week 12: Pain vs. PGA | 0.612 [0.562 to 0.657]
  Week 12: PHQ-2 vs. PGA: number analyzed (Participants) | 728
  Week 12: PHQ-2 vs. PGA | 0.376 [0.312 to 0.436]
  Week 24: PtGA vs. Fatigue: number analyzed (Participants) | 588
  Week 24: PtGA vs. Fatigue | 0.588 [0.532 to 0.638]
  Week 24: PtGA vs. Pain: number analyzed (Participants) | 593
  Week 24: PtGA vs. Pain | 0.859 [0.837 to 0.879]
  Week 24: PtGA vs. PHQ-2: number analyzed (Participants) | 593
  Week 24: PtGA vs. PHQ-2 | 0.526 [0.465 to 0.582]
  Week 24: PtGA vs. PGA: number analyzed (Participants) | 580
  Week 24: PtGA vs. PGA | 0.600 [0.545 to 0.650]
  Week 24: Fatigue vs. Pain: number analyzed (Participants) | 585
  Week 24: Fatigue vs. Pain | 0.621 [0.569 to 0.668]
  Week 24: Fatigue vs. PHQ-2: number analyzed (Participants) | 586
  Week 24: Fatigue vs. PHQ-2 | 0.591 [0.536 to 0.641]
  Week 24: Fatigue vs. PGA: number analyzed (Participants) | 571
  Week 24: Fatigue vs. PGA | 0.389 [0.317 to 0.456]
  Week 24: Pain vs. PHQ-2: number analyzed (Participants) | 589
  Week 24: Pain vs. PHQ-2 | 0.558 [0.500 to 0.611]
  Week 24: Pain vs. PGA: number analyzed (Participants) | 576
  Week 24: Pain vs. PGA | 0.556 [0.497 to 0.610]
  Week 24: PHQ-2 vs. PGA: number analyzed (Participants) | 611
  Week 24: PHQ-2 vs. PGA | 0.379 [0.309 to 0.445]
  Week 36: PtGA vs. Fatigue: number analyzed (Participants) | 503
  Week 36: PtGA vs. Fatigue | 0.664 [0.611 to 0.710]
  Week 36: PtGA vs. Pain: number analyzed (Participants) | 501
  Week 36: PtGA vs. Pain | 0.839 [0.810 to 0.863]
  Week 36: PtGA vs. PHQ-2: number analyzed (Participants) | 505
  Week 36: PtGA vs. PHQ-2 | 0.513 [0.445 to 0.574]
  Week 36: PtGA vs. PGA: number analyzed (Participants) | 499
  Week 36: PtGA vs. PGA | 0.609 [0.550 to 0.661]
  Week 36: Fatigue vs. Pain: number analyzed (Participants) | 500
  Week 36: Fatigue vs. Pain | 0.646 [0.591 to 0.694]
  Week 36: Fatigue vs. PHQ-2: number analyzed (Participants) | 505
  Week 36: Fatigue vs. PHQ-2 | 0.614 [0.556 to 0.665]
  Week 36: Fatigue vs. PGA: number analyzed (Participants) | 499
  Week 36: Fatigue vs. PGA | 0.463 [0.391 to 0.529]
  Week 36: Pain vs. PHQ-2: number analyzed (Participants) | 501
  Week 36: Pain vs. PHQ-2 | 0.532 [0.466 to 0.592]
  Week 36: Pain vs. PGA: number analyzed (Participants) | 495
  Week 36: Pain vs. PGA | 0.576 [0.514 to 0.632]
  Week 36: PHQ-2 vs. PGA: number analyzed (Participants) | 530
  Week 36: PHQ-2 vs. PGA | 0.367 [0.291 to 0.438]
  Week 52: PtGA vs. Fatigue: number analyzed (Participants) | 434
  Week 52: PtGA vs. Fatigue | 0.666 [0.609 to 0.715]
  Week 52: PtGA vs. Pain: number analyzed (Participants) | 439
  Week 52: PtGA vs. Pain | 0.861 [0.835 to 0.884]
  Week 52: PtGA vs. PHQ-2: number analyzed (Participants) | 437
  Week 52: PtGA vs. PHQ-2 | 0.507 [0.434 to 0.574]
  Week 52: PtGA vs. PGA: number analyzed (Participants) | 434
  Week 52: PtGA vs. PGA | 0.632 [0.571 to 0.685]
  Week 52: Fatigue vs. Pain: number analyzed (Participants) | 433
  Week 52: Fatigue vs. Pain | 0.649 [0.591 to 0.700]
  Week 52: Fatigue vs. PHQ-2: number analyzed (Participants) | 433
  Week 52: Fatigue vs. PHQ-2 | 0.574 [0.507 to 0.633]
  Week 52: Fatigue vs. PGA: number analyzed (Participants) | 429
  Week 52: Fatigue vs. PGA | 0.485 [0.409 to 0.554]
  Week 52: Pain vs. PHQ-2: number analyzed (Participants) | 435
  Week 52: Pain vs. PHQ-2 | 0.545 [0.475 to 0.607]
  Week 52: Pain vs. PGA: number analyzed (Participants) | 432
  Week 52: Pain vs. PGA | 0.641 [0.582 to 0.693]
  Week 52: PHQ-2 vs. PGA: number analyzed (Participants) | 454
  Week 52: PHQ-2 vs. PGA | 0.445 [0.367 to 0.515]

22. Secondary Outcome: Ankylosing Spondylitis (axSpA): Spearman Correlation Coefficient Between Patient Global Assessment (PtGA) of Disease Activity, VAS Fatigue, VAS Pain Score, Patient Health Quessionare-2 (PHQ-2) and PGA of Disease Activity at Weeks 12, 24, 36, 52
Description: as for outcome 21
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with axSpA. "Number analyzed" signifies participants analyzed for this outcome measure at specified time points.
Measure: Number (95% Confidence Interval); unit: spearman correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 305
spearman correlation coefficient
  Week 12:PtGA vs. Fatigue: number analyzed (Participants) | 247
  Week 12:PtGA vs. Fatigue | 0.582 [0.492 to 0.658]
  Week 12: PtGA vs. Pain: number analyzed (Participants) | 246
  Week 12: PtGA vs. Pain | 0.899 [0.872 to 0.921]
  Week 12: PtGA vs. PHQ-2: number analyzed (Participants) | 242
  Week 12: PtGA vs. PHQ-2 | 0.526 [0.427 to 0.611]
  Week 12: PtGA vs. PGA: number analyzed (Participants) | 247
  Week 12: PtGA vs. PGA | 0.606 [0.520 to 0.679]
  Week 12: Fatigue vs. Pain: number analyzed (Participants) | 251
  Week 12: Fatigue vs. Pain | 0.547 [0.453 to 0.628]
  Week 12: Fatigue vs. PHQ-2: number analyzed (Participants) | 248
  Week 12: Fatigue vs. PHQ-2 | 0.487 [0.384 to 0.576]
  Week 12: Fatigue vs. PGA: number analyzed (Participants) | 253
  Week 12: Fatigue vs. PGA | 0.369 [0.256 to 0.470]
  Week 12: Pain vs. PHQ-2: number analyzed (Participants) | 245
  Week 12: Pain vs. PHQ-2 | 0.530 [0.433 to 0.614]
  Week 12: Pain vs. PGA: number analyzed (Participants) | 250
  Week 12: Pain vs. PGA | 0.617 [0.533 to 0.688]
  Week 12: PHQ-2 vs. PGA: number analyzed (Participants) | 269
  Week 12: PHQ-2 vs. PGA | 0.392 [0.285 to 0.488]
  Week 24: PtGA vs. Fatigue: number analyzed (Participants) | 204
  Week 24: PtGA vs. Fatigue | 0.668 [0.584 to 0.737]
  Week 24: PtGA vs. Pain: number analyzed (Participants) | 206
  Week 24: PtGA vs. Pain | 0.904 [0.874 to 0.926]
  Week 24: PtGA vs. PHQ-2: number analyzed (Participants) | 205
  Week 24: PtGA vs. PHQ-2 | 0.495 [0.383 to 0.591]
  Week 24: PtGA vs. PGA: number analyzed (Participants) | 205
  Week 24: PtGA vs. PGA | 0.495 [0.383 to 0.591]
  Week 24: Fatigue vs. Pain: number analyzed (Participants) | 204
  Week 24: Fatigue vs. Pain | 0.664 [0.578 to 0.734]
  Week 24: Fatigue vs. PHQ-2: number analyzed (Participants) | 203
  Week 24: Fatigue vs. PHQ-2 | 0.634 [0.543 to 0.709]
  Week 24: Fatigue vs. PGA: number analyzed (Participants) | 204
  Week 24: Fatigue vs. PGA | 0.445 [0.326 to 0.548]
  Week 24: Pain vs. PHQ-2: number analyzed (Participants) | 205
  Week 24: Pain vs. PHQ-2 | 0.492 [0.379 to 0.588]
  Week 24: Pain vs. PGA: number analyzed (Participants) | 205
  Week 24: Pain vs. PGA | 0.515 [0.405 to 0.608]
  Week 24: PHQ-2 vs. PGA: number analyzed (Participants) | 215
  Week 24: PHQ-2 vs. PGA | 0.449 [0.335 to 0.549]
  Week 36: PtGA vs. Fatigue: number analyzed (Participants) | 183
  Week 36: PtGA vs. Fatigue | 0.720 [0.641 to 0.782]
  Week 36: PtGA vs. Pain: number analyzed (Participants) | 184
  Week 36: PtGA vs. Pain | 0.914 [0.886 to 0.935]
  Week 36: PtGA vs. PHQ-2: number analyzed (Participants) | 184
  Week 36: PtGA vs. PHQ-2 | 0.630 [0.533 to 0.709]
  Week 36: PtGA vs. PGA: number analyzed (Participants) | 185
  Week 36: PtGA vs. PGA | 0.586 [0.481 to 0.672]
  Week 36: Fatigue vs. Pain: number analyzed (Participants) | 181
  Week 36: Fatigue vs. Pain | 0.728 [0.650 to 0.789]
  Week 36: Fatigue vs. PHQ-2: number analyzed (Participants) | 182
  Week 36: Fatigue vs. PHQ-2 | 0.691 [0.606 to 0.759]
  Week 36: Fatigue vs. PGA: number analyzed (Participants) | 183
  Week 36: Fatigue vs. PGA | 0.530 [0.415 to 0.626]
  Week 36: Pain vs. PHQ-2: number analyzed (Participants) | 183
  Week 36: Pain vs. PHQ-2 | 0.637 [0.540 to 0.715]
  Week 36: Pain vs. PGA: number analyzed (Participants) | 184
  Week 36: Pain vs. PGA | 0.591 [0.487 to 0.677]
  Week 36: PHQ-2 vs. PGA: number analyzed (Participants) | 195
  Week 36: PHQ-2 vs. PGA | 0.483 [0.366 to 0.583]
  Week 52: PtGA vs. Fatigue: number analyzed (Participants) | 171
  Week 52: PtGA vs. Fatigue | 0.717 [0.634 to 0.782]
  Week 52: PtGA vs. Pain: number analyzed (Participants) | 172
  Week 52: PtGA vs. Pain | 0.912 [0.882 to 0.934]
  Week 52: PtGA vs. PHQ-2: number analyzed (Participants) | 170
  Week 52: PtGA vs. PHQ-2 | 0.586 [0.476 to 0.676]
  Week 52: PtGA vs. PGA: number analyzed (Participants) | 171
  Week 52: PtGA vs. PGA | 0.548 [0.432 to 0.644]
  Week 52: Fatigue vs. Pain: number analyzed (Participants) | 171
  Week 52: Fatigue vs. Pain | 0.743 [0.666 to 0.803]
  Week 52: Fatigue vs. PHQ-2: number analyzed (Participants) | 172
  Week 52: Fatigue vs. PHQ-2 | 0.676 [0.584 to 0.749]
  Week 52: Fatigue vs. PGA: number analyzed (Participants) | 171
  Week 52: Fatigue vs. PGA | 0.457 [0.328 to 0.567]
  Week 52: Pain vs. PHQ-2: number analyzed (Participants) | 170
  Week 52: Pain vs. PHQ-2 | 0.629 [0.527 to 0.711]
  Week 52: Pain vs. PGA: number analyzed (Participants) | 171
  Week 52: Pain vs. PGA | 0.603 [0.497 to 0.690]
  Week 52: PHQ-2 vs. PGA: number analyzed (Participants) | 179
  Week 52: PHQ-2 vs. PGA | 0.420 [0.290 to 0.533]

23. Secondary Outcome: Psoriatic Arthritis (PsA): Spearman Correlation Coefficient Between Patient Global Assessment (PtGA) of Disease Activity, VAS Fatigue, VAS Pain Score, Patient Health Quessionare-2 (PHQ-2) and PGA of Disease Activity at Weeks 12, 24, 36, 52
Description: as for outcome 21
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with PsA. Number analyzed signifies participants analyzed for this outcome measure at specified time points.
Measure: Number (95% Confidence Interval); unit: spearman correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 254
spearman correlation coefficient
  Week 12: PtGA vs. Fatigue: number analyzed (Participants) | 220
  Week 12: PtGA vs. Fatigue | 0.630 [0.542 to 0.703]
  Week 12: PtGA vs. Pain: number analyzed (Participants) | 222
  Week 12: PtGA vs. Pain | 0.892 [0.862 to 0.916]
  Week 12: PtGA vs. PHQ-2: number analyzed (Participants) | 219
  Week 12: PtGA vs. PHQ-2 | 0.609 [0.518 to 0.686]
  Week 12: PtGA vs. PGA: number analyzed (Participants) | 215
  Week 12: PtGA vs. PGA | 0.509 [0.402 to 0.601]
  Week 12: Fatigue vs. Pain: number analyzed (Participants) | 222
  Week 12: Fatigue vs. Pain | 0.664 [0.583 to 0.731]
  Week 12: Fatigue vs. PHQ-2: number analyzed (Participants) | 220
  Week 12: Fatigue vs. PHQ-2 | 0.601 [0.508 to 0.678]
  Week 12: Fatigue vs. PGA: number analyzed (Participants) | 215
  Week 12: Fatigue vs. PGA | 0.324 [0.198 to 0.438]
  Week 12: Pain vs. PHQ-2: number analyzed (Participants) | 221
  Week 12: Pain vs. PHQ-2 | 0.628 [0.540 to 0.701]
  Week 12: Pain vs. PGA: number analyzed (Participants) | 217
  Week 12: Pain vs. PGA | 0.529 [0.425 to 0.618]
  Week 12: PHQ-2 vs. PGA: number analyzed (Participants) | 223
  Week 12: PHQ-2 vs. PGA | 0.381 [0.262 to 0.488]
  Week 24: PtGA vs. Fatigue: number analyzed (Participants) | 187
  Week 24: PtGA vs. Fatigue | 0.656 [0.565 to 0.730]
  Week 24: PtGA vs. Pain: number analyzed (Participants) | 190
  Week 24: PtGA vs. Pain | 0.881 [0.844 to 0.909]
  Week 24: PtGA vs. PHQ-2: number analyzed (Participants) | 187
  Week 24: PtGA vs. PHQ-2 | 0.562 [0.454 to 0.652]
  Week 24: PtGA vs. PGA: number analyzed (Participants) | 189
  Week 24: PtGA vs. PGA | 0.559 [0.451 to 0.649]
  Week 24: Fatigue vs. Pain: number analyzed (Participants) | 188
  Week 24: Fatigue vs. Pain | 0.674 [0.586 to 0.744]
  Week 24: Fatigue vs. PHQ-2: number analyzed (Participants) | 187
  Week 24: Fatigue vs. PHQ-2 | 0.620 [0.521 to 0.700]
  Week 24: Fatigue vs. PGA: number analyzed (Participants) | 188
  Week 24: Fatigue vs. PGA | 0.374 [0.243 to 0.490]
  Week 24: Pain vs. PHQ-2: number analyzed (Participants) | 188
  Week 24: Pain vs. PHQ-2 | 0.607 [0.507 to 0.690]
  Week 24: Pain vs. PGA: number analyzed (Participants) | 190
  Week 24: Pain vs. PGA | 0.630 [0.534 to 0.708]
  Week 24: PHQ-2 vs. PGA: number analyzed (Participants) | 195
  Week 24: PHQ-2 vs. PGA | 0.410 [0.285 to 0.520]
  Week 36: PtGA vs. Fatigue: number analyzed (Participants) | 170
  Week 36: PtGA vs. Fatigue | 0.692 [0.603 to 0.762]
  Week 36: PtGA vs. Pain: number analyzed (Participants) | 173
  Week 36: PtGA vs. Pain | 0.913 [0.884 to 0.935]
  Week 36: PtGA vs. PHQ-2: number analyzed (Participants) | 170
  Week 36: PtGA vs. PHQ-2 | 0.645 [0.546 to 0.724]
  Week 36: PtGA vs. PGA: number analyzed (Participants) | 172
  Week 36: PtGA vs. PGA | 0.513 [0.392 to 0.614]
  Week 36: Fatigue vs. Pain: number analyzed (Participants) | 169
  Week 36: Fatigue vs. Pain | 0.724 [0.642 to 0.788]
  Week 36: Fatigue vs. PHQ-2: number analyzed (Participants) | 168
  Week 36: Fatigue vs. PHQ-2 | 0.710 [0.624 to 0.777]
  Week 36: Fatigue vs. PGA: number analyzed (Participants) | 169
  Week 36: Fatigue vs. PGA | 0.423 [0.290 to 0.539]
  Week 36: Pain vs. PHQ-2: number analyzed (Participants) | 169
  Week 36: Pain vs. PHQ-2 | 0.658 [0.561 to 0.735]
  Week 36: Pain vs. PGA: number analyzed (Participants) | 171
  Week 36: Pain vs. PGA | 0.532 [0.414 to 0.631]
  Week 36: PHQ-2 vs. PGA: number analyzed (Participants) | 172
  Week 36: PHQ-2 vs. PGA | 0.357 [0.218 to 0.480]
  Week 52: PtGA vs. Fatigue: number analyzed (Participants) | 144
  Week 52: PtGA vs. Fatigue | 0.753 [0.671 to 0.815]
  Week 52: PtGA vs. Pain: number analyzed (Participants) | 144
  Week 52: PtGA vs. Pain | 0.908 [0.874 to 0.933]
  Week 52: PtGA vs. PHQ-2: number analyzed (Participants) | 144
  Week 52: PtGA vs. PHQ-2 | 0.696 [0.599 to 0.771]
  Week 52: PtGA vs. PGA: number analyzed (Participants) | 142
  Week 52: PtGA vs. PGA | 0.565 [0.439 to 0.666]
  Week 52: Fatigue vs. Pain: number analyzed (Participants) | 146
  Week 52: Fatigue vs. Pain | 0.760 [0.680 to 0.820]
  Week 52: Fatigue vs. PHQ-2: number analyzed (Participants) | 145
  Week 52: Fatigue vs. PHQ-2 | 0.726 [0.637 to 0.794]
  Week 52: Fatigue vs. PGA: number analyzed (Participants) | 144
  Week 52: Fatigue vs. PGA | 0.430 [0.285 to 0.553]
  Week 52: Pain vs. PHQ-2: number analyzed (Participants) | 145
  Week 52: Pain vs. PHQ-2 | 0.683 [0.584 to 0.761]
  Week 52: Pain vs. PGA: number analyzed (Participants) | 144
  Week 52: Pain vs. PGA | 0.581 [0.459 to 0.679]
  Week 52: PHQ-2 vs. PGA: number analyzed (Participants) | 147
  Week 52: PHQ-2 vs. PGA | 0.498 [0.364 to 0.609]

24. Secondary Outcome: Plaque Psoriasis (PsO): Spearman Correlation Coefficient Between Patient Global Assessment (PtGA) of Disease Activity, VAS Fatigue, VAS Pain Score, Patient Health Quessionare-2 (PHQ-2) and PGA of Disease Activity at Weeks 12, 24, 36, 52
Description: as for outcome 21
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with PsO. "Number analyzed" signifies participants analyzed for this outcome measure at specified time points.
Measure: Number (95% Confidence Interval); unit: spearman correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 70
spearman correlation coefficient
  Week 12: PtGA vs. Fatigue: number analyzed (Participants) | 62
  Week 12: PtGA vs. Fatigue | 0.350 [0.107 to 0.550]
  Week 12: PtGA vs. Pain: number analyzed (Participants) | 61
  Week 12: PtGA vs. Pain | 0.606 [0.414 to 0.742]
  Week 12: PtGA vs. PHQ-2: number analyzed (Participants) | 58
  Week 12: PtGA vs. PHQ-2 | 0.563 [0.353 to 0.715]
  Week 12: PtGA vs. PGA: number analyzed (Participants) | 62
  Week 12: PtGA vs. PGA | 0.606 [0.415 to 0.741]
  Week 12: Fatigue vs. Pain: number analyzed (Participants) | 63
  Week 12: Fatigue vs. Pain | 0.679 [0.515 to 0.791]
  Week 12: Fatigue vs. PHQ-2: number analyzed (Participants) | 60
  Week 12: Fatigue vs. PHQ-2 | 0.681 [0.512 to 0.795]
  Week 12: Fatigue vs. PGA: number analyzed (Participants) | 64
  Week 12: Fatigue vs. PGA | 0.175 [-0.075 to 0.403]
  Week 12: Pain vs. PHQ-2: number analyzed (Participants) | 59
  Week 12: Pain vs. PHQ-2 | 0.647 [0.464 to 0.772]
  Week 12: Pain vs. PGA: number analyzed (Participants) | 63
  Week 12: Pain vs. PGA | 0.384 [0.147 to 0.575]
  Week 12: PHQ-2 vs. PGA: number analyzed (Participants) | 63
  Week 12: PHQ-2 vs. PGA | 0.265 [0.016 to 0.479]
  Week 24: PtGA vs. Fatigue: number analyzed (Participants) | 50
  Week 24: PtGA vs. Fatigue | 0.651 [0.450 to 0.784]
  Week 24: PtGA vs. Pain: number analyzed (Participants) | 50
  Week 24: PtGA vs. Pain | 0.692 [0.508 to 0.812]
  Week 24: PtGA vs. PHQ-2: number analyzed (Participants) | 49
  Week 24: PtGA vs. PHQ-2 | 0.485 [0.231 to 0.672]
  Week 24: PtGA vs. PGA: number analyzed (Participants) | 50
  Week 24: PtGA vs. PGA | 0.713 [0.537 to 0.825]
  Week 24: Fatigue vs. Pain: number analyzed (Participants) | 50
  Week 24: Fatigue vs. Pain | 0.802 [0.669 to 0.881]
  Week 24: Fatigue vs. PHQ-2: number analyzed (Participants) | 49
  Week 24: Fatigue vs. PHQ-2 | 0.577 [0.348 to 0.736]
  Week 24: Fatigue vs. PGA: number analyzed (Participants) | 50
  Week 24: Fatigue vs. PGA | 0.377 [0.107 to 0.591]
  Week 24: Pain vs. PHQ-2: number analyzed (Participants) | 49
  Week 24: Pain vs. PHQ-2 | 0.466 [0.208 to 0.658]
  Week 24: Pain vs. PGA: number analyzed (Participants) | 50
  Week 24: Pain vs. PGA | 0.470 [0.216 to 0.659]
  Week 24: PHQ-2 vs. PGA: number analyzed (Participants) | 51
  Week 24: PHQ-2 vs. PGA | 0.219 [-0.062 to 0.465]
  Week 36: PtGA vs. Fatigue: number analyzed (Participants) | 38
  Week 36: PtGA vs. Fatigue | 0.627 [0.377 to 0.785]
  Week 36: PtGA vs. Pain: number analyzed (Participants) | 38
  Week 36: PtGA vs. Pain | 0.687 [0.463 to 0.822]
  Week 36: PtGA vs. PHQ-2: number analyzed (Participants) | 38
  Week 36: PtGA vs. PHQ-2 | 0.585 [0.319 to 0.759]
  Week 36: PtGA vs. PGA: number analyzed (Participants) | 38
  Week 36: PtGA vs. PGA | 0.519 [0.233 to 0.716]
  Week 36: Fatigue vs. Pain: number analyzed (Participants) | 39
  Week 36: Fatigue vs. Pain | 0.744 [0.553 to 0.855]
  Week 36: Fatigue vs. PHQ-2: number analyzed (Participants) | 39
  Week 36: Fatigue vs. PHQ-2 | 0.812 [0.661 to 0.895]
  Week 36: Fatigue vs. PGA: number analyzed (Participants) | 39
  Week 36: Fatigue vs. PGA | 0.288 [-0.034 to 0.550]
  Week 36: Pain vs. PHQ-2: number analyzed (Participants) | 39
  Week 36: Pain vs. PHQ-2 | 0.659 [0.426 to 0.803]
  Week 36: Pain vs. PGA: number analyzed (Participants) | 39
  Week 36: Pain vs. PGA | 0.411 [0.104 to 0.640]
  Week 36: PHQ-2 vs. PGA: number analyzed (Participants) | 41
  Week 36: PHQ-2 vs. PGA | 0.167 [-0.150 to 0.450]
  Week 52: PtGA vs. Fatigue: number analyzed (Participants) | 32
  Week 52: PtGA vs. Fatigue | 0.418 [0.074 to 0.665]
  Week 52: PtGA vs. Pain: number analyzed (Participants) | 33
  Week 52: PtGA vs. Pain | 0.625 [0.350 to 0.794]
  Week 52: PtGA vs. PHQ-2: number analyzed (Participants) | 33
  Week 52: PtGA vs. PHQ-2 | 0.464 [0.137 to 0.693]
  Week 52: PtGA vs. PGA: number analyzed (Participants) | 33
  Week 52: PtGA vs. PGA | 0.753 [0.544 to 0.868]
  Week 52: Fatigue vs. Pain: number analyzed (Participants) | 32
  Week 52: Fatigue vs. Pain | 0.579 [0.281 to 0.768]
  Week 52: Fatigue vs. PHQ-2: number analyzed (Participants) | 32
  Week 52: Fatigue vs. PHQ-2 | 0.598 [0.307 to 0.780]
  Week 52: Fatigue vs. PGA: number analyzed (Participants) | 32
  Week 52: Fatigue vs. PGA | 0.278 [-0.083 to 0.568]
  Week 52: Pain vs. PHQ-2: number analyzed (Participants) | 33
  Week 52: Pain vs. PHQ-2 | 0.404 [0.064 to 0.653]
  Week 52: Pain vs. PGA: number analyzed (Participants) | 33
  Week 52: Pain vs. PGA | 0.421 [0.085 to 0.664]
  Week 52: PHQ-2 vs. PGA: number analyzed (Participants) | 36
  Week 52: PHQ-2 vs. PGA | 0.208 [-0.132 to 0.500]

25. Secondary Outcome: Rheumatoid Arthritis(RA): Spearman Correlation Coefficient Between Hannover Functional Questionnaire (FFbH) and Morning Stiffness at Weeks 12, 24, 36, 52
Description: FFbH consists 18 questions to assess daily activities in last 7 days. Each question is answered by the participant as "Yes, I can perform the activity without difficulty" (score assigned = 2), "Yes, but with some difficulties" (score assigned = 1) and "No or only with help" (score assigned = 0). Final FFbH score (FFbH functional capacity) was then computed according to formula: (Sum of all single scores * 100% [percent]) / (2 * number of answered questions) ranged between 0-100; higher score indicates better daily activities. Duration of morning stiffness was defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes (If none was present = 0; If morning stiffness was continuing at the time of assessment or was unusual compared to the recent past, average of duration of stiffness over the past 3 days was reported; If stiffness persisted the entire day, 1440 minutes [24 hours*60 minutes] was recorded).
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: spearman correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 824
spearman correlation coefficient
  Week 12: FFbH vs. Morning stiffness: number analyzed (Participants) | 661
  Week 12: FFbH vs. Morning stiffness | -0.439 [-0.498 to -0.375]
  Week 24: FFbH vs. Morning stiffness: number analyzed (Participants) | 560
  Week 24: FFbH vs. Morning stiffness | -0.486 [-0.547 to -0.420]
  Week 36: FFbH vs. Morning stiffness: number analyzed (Participants) | 477
  Week 36: FFbH vs. Morning stiffness | -0.520 [-0.582 to -0.451]
  Week 52: FFbH vs. Morning stiffness: number analyzed (Participants) | 417
  Week 52: FFbH vs. Morning stiffness | -0.502 [-0.571 to -0.427]

26. Secondary Outcome: Psoriatic Arthritis(PsA): Spearman Correlation Coefficient Between Hannover Functional Questionnaire (FFbH) and Morning Stiffness at Weeks 12, 24, 36, 52
Description: as for outcome 25
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with PsA. "Number analyzed" signifies participants analyzed for this outcome measure at specified time points.
Measure: Number (95% Confidence Interval); unit: spearman correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 254
spearman correlation coefficient
  Week 12: FFbH vs. Morning stiffness: number analyzed (Participants) | 206
  Week 12: FFbH vs. Morning stiffness | -0.493 [-0.589 to -0.381]
  Week 24: FFbH vs. Morning stiffness: number analyzed (Participants) | 175
  Week 24: FFbH vs. Morning stiffness | -0.640 [-0.719 to -0.542]
  Week 36: FFbH vs. Morning stiffness: number analyzed (Participants) | 154
  Week 36: FFbH vs. Morning stiffness | -0.615 [-0.703 to -0.504]
  Week 52: FFbH vs. Morning stiffness: number analyzed (Participants) | 130
  Week 52: FFbH vs. Morning stiffness | -0.560 [-0.667 to -0.428]

27. Secondary Outcome: Ankylosing Spondylitis(axSpA): Spearman Correlation Coefficient Between Hannover Functional Questionnaire (FFbH) and Morning Stiffness at Weeks 12, 24, 36, 52
Description: as for outcome 25
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: spearman correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 305
spearman correlation coefficient
  Week 12: FFbH vs. Morning stiffness: number analyzed (Participants) | 245
  Week 12: FFbH vs. Morning stiffness | -0.523 [-0.608 to -0.425]
  Week 24: FFbH vs. Morning stiffness: number analyzed (Participants) | 198
  Week 24: FFbH vs. Morning stiffness | -0.523 [-0.617 to -0.413]
  Week 36: FFbH vs. Morning stiffness: number analyzed (Participants) | 172
  Week 36: FFbH vs. Morning stiffness | -0.565 [-0.658 to -0.453]
  Week 52: FFbH vs. Morning stiffness: number analyzed (Participants) | 159
  Week 52: FFbH vs. Morning stiffness | -0.600 [-0.690 to -0.489]

28. Secondary Outcome: Percentage of Participants Who Discontinued Treatment Due to Lack of Efficacy or Adverse Events
Description: Percentage of participants who discontinued etanercept before completing the study, was reported.
Time Frame: Baseline up to Week 52
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1465
percentage of participants
  Due to lack of Efficacy | 15.2
  Due to Adverse Events | 8.5

29. Secondary Outcome: Number of Participants Who Switched to Other Therapy After Treatment Discontinuation
Description: Participants who switched from etanercept to either disease-modifying antirheumatic drugs (DMARDs) or alternative biologic drug were reported.
Time Frame: Baseline up to Week 52
Population: Treated set included all documented participants who were treated, had at least 1 post-baseline value and had an AE documented. Overall number of participants analyzed signifies participants from treated set who discontinued treatment with Etanercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 410
Participants
  Abatacept | 15
  Adalimumab | 53
  Apremilast | 7
  Azathioprin | 1
  Azathioprin, Leflunomid, Diclofenac | 1
  Azathioprin, Prednisolon | 1
  Baricitinib | 3
  Biological NOS | 5
  Certolizumab | 26
  Etanercept Biosimilar | 10
  Golimumab | 6
  Hydroxychloroquin | 1
  Leflunomid | 4
  Methotrexate (MTX) | 6
  MTX, Adalimumab | 2
  MTX, Prednisolon | 3
  MTX, Tocilizumab | 1
  Prednisolon | 13
  Prednisolon, Diclofenac | 1
  Remsima (Infliximab-Biosimilar) | 1
  Rituximab | 12
  Roactemra | 10
  Secukinumab | 27
  Sulfasalazin | 1
  Sulfasalazin, Leflunomid | 1
  Tapentadol | 2
  Tocilizumab | 25
  Tofacitinib | 2
  Ustekinumab | 7
  Etoricoxib | 1
  Ibuprofen | 2
  Ibuprofen, Metamizol | 1
  Ibuprofen, Prednisolon, Oxycodon, Pregabalin | 1
  Inflectra (Infliximab Biosimilar) | 1
  Infliximab | 1
  NSAR | 1
  Corticosteroid | 1
  PUVA | 1
  Unknown | 5
  None | 56
  Missing values | 92

30. Secondary Outcome: Hannover Functional Questionnaire (FFbH) Functional Capacity Score of Participants With Rheumatoid Arthritis (RA), Axial Spondyloarthritis (axSpA), Psoriasis Arthritis (PsA) at Weeks 12, 24, 36, 52
Description: FFbH consisted 18 questions to assess daily activities in last 7 days. Each question was answered by the participant as "Yes, I can perform the activity without difficulty" (score assigned = 2), "Yes, but with some difficulties" (score assigned = 1) and "No or only with help" (score assigned = 0). Final FFbH score (FFbH functional capacity) was then computed according to formula: (Sum of all single scores * 100% [percent]) / (2 * number of answered questions) ranged between 0-100; higher score indicated better daily activities.
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with RA, axSpA or PsA. "Number analyzed" signifies participants analyzed for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Etanercept: All participants with RA, axSpA or PsA taking etanercept in the routine treatment as per clinical practice and in line with summary of product characteristics clinical, were observed for a period of 12 months.
Arm/Group | Etanercept
Number analyzed (Participants) | 1383
units on a scale
  Week 12: number analyzed (Participants) | 1264
  Week 12 | 71.4 (22.2)
  Week 24: number analyzed (Participants) | 1068
  Week 24 | 72.2 (22.4)
  Week 36: number analyzed (Participants) | 915
  Week 36 | 73.4 (22.3)
  Week 52: number analyzed (Participants) | 803
  Week 52 | 73.7 (22.5)

31. Secondary Outcome: Clinical Disease Activity Index (CDAI) Scores of Participants With Rheumatoid Arthritis (RA) at Weeks 12, 24, 36 and 52
Description: The CDAI is the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and PGA assessed on 0-10 cm VAS; higher scores=greater affection due to disease activity. CDAI total score = 0-76. CDAI <= 2.8 indicates disease remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high disease activity.
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 824
units on a scale
  Week 12: number analyzed (Participants) | 668
  Week 12 | 12.7 (9.7)
  Week 24: number analyzed (Participants) | 572
  Week 24 | 11.0 (9.4)
  Week 36: number analyzed (Participants) | 496
  Week 36 | 10.1 (8.9)
  Week 52: number analyzed (Participants) | 433
  Week 52 | 9.2 (9.1)

32. Secondary Outcome: Simplified Disease Activity Index (SDAI) Scores of Participants With Rheumatoid Arthritis (RA) at Weeks 12, 24, 36 and 52
Description: The SDAI is the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and PGA assessed on 0-10 cm VAS; higher scores=greater affection due to disease activity, and C-reactive protein (CRP) (mg/dL). SDAI total score= 0-86. SDAI <=3.3 indicates disease remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high disease activity.
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 824
units on a scale
  Week 12: number analyzed (Participants) | 594
  Week 12 | 14.3 (11.0)
  Week 24: number analyzed (Participants) | 494
  Week 24 | 12.0 (11.3)
  Week 36: number analyzed (Participants) | 428
  Week 36 | 11.1 (9.7)
  Week 52: number analyzed (Participants) | 379
  Week 52 | 10.1 (10.2)

33. Secondary Outcome: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) of Participants With Axial Spondyloarthritis (axSpA) at Weeks 12, 24, 36 and 52
Description: BASDAI is a validated self-assessment tool used to determine disease activity in participant with ankylosing spondylitis. Utilizing a VAS of 0-10 (0=none and 10=very severe) participant's answered 6 questions measuring discomfort, pain and fatigue. The final BASDAI score averages the individual assessments for a final score range of 0(no symptoms)-10(very severe symptoms).
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 305
units on a scale
  Week 12: number analyzed (Participants) | 265
  Week 12 | 3.8 (2.3)
  Week 24: number analyzed (Participants) | 209
  Week 24 | 3.5 (2.3)
  Week 36: number analyzed (Participants) | 190
  Week 36 | 3.2 (2.1)
  Week 52: number analyzed (Participants) | 182
  Week 52 | 3.3 (2.2)

34. Secondary Outcome: Number of Affected Enthesis in Participants With Axial Spondyloarthritis (axSpA) and Psoriatic Arthritis(PsA) at Weeks 12, 24, 36 and 52
Description: An enthesis is the site where the joint capsules, ligaments or tendons attach to the bone. Enthesitis is the inflammation of the entheses. This inflammation can lead to severe pain and discomfort.
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with axSpA or PsA. "Number analyzed" signifies participants analyzed for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: enthesis
Groups:
- Etanercept: All participants with axSpA or PsA taking etanercept in the routine treatment as per clinical practice and in line with summary of product characteristics clinical, were observed for a period of 12 months.
Arm/Group | Etanercept
Number analyzed (Participants) | 559
enthesis
  Week 12: number analyzed (Participants) | 90
  Week 12 | 1.0 (1.8)
  Week 24: number analyzed (Participants) | 78
  Week 24 | 0.6 (1.2)
  Week 36: number analyzed (Participants) | 66
  Week 36 | 0.4 (1.1)
  Week 52: number analyzed (Participants) | 60
  Week 52 | 0.3 (1.0)

35. Secondary Outcome: Occiput-to-wall Distance of Participants With Axial Spondyloarthritis (axSpA) at Weeks 12, 24, 36 and 52
Description: Occiput-to-wall distance was the distance between the occiput (posterior or back portion of the head) and the wall when the participant stood with heels and shoulder against the wall and the back straight.
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 305
cm
  Week 12: number analyzed (Participants) | 227
  Week 12 | 6.7 (10.7)
  Week 24: number analyzed (Participants) | 184
  Week 24 | 6.6 (11.3)
  Week 36: number analyzed (Participants) | 166
  Week 36 | 6.3 (11.2)
  Week 52: number analyzed (Participants) | 150
  Week 52 | 6.0 (11.0)

36. Secondary Outcome: Mean Percentage of Total Body Surface Area (BSA) for Participants With Plaque Psoriasis (PsO) and Psoriasis Arthritis (PsA) at Weeks 12, 24, 36 and 52
Description: Percentage of BSA affected by psoriasis was estimated using the palm method: one of the participant's palm to proximal interphalangeal and thumb = 1 percent (%) of total BSA. Regions of the body were assigned specific number of palms with percentage [Head and neck = 10% (10 palms), upper extremities = 20% (20 palms), Trunk (axillae and groin) = 30% (30 palms), lower extremities (buttocks) = 40% (40 palms)]. The total BSA affected was the summation of individual regions affected.
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with PsO, PsA. "Number analyzed" signifies participants analyzed for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: percentage of BSA
Groups:
- Etanercept: All participants with PsO, PsA taking etanercept in the routine treatment as per clinical practice and in line with summary of product characteristics clinical, were observed for a period of 12 months.
Arm/Group | Etanercept
Number analyzed (Participants) | 324
percentage of BSA
  Week 12: number analyzed (Participants) | 245
  Week 12 | 8.5 (12.8)
  Week 24: number analyzed (Participants) | 205
  Week 24 | 5.9 (9.2)
  Week 36: number analyzed (Participants) | 176
  Week 36 | 4.8 (7.1)
  Week 52: number analyzed (Participants) | 162
  Week 52 | 5.4 (10.9)

37. Secondary Outcome: Mean of Total Number of Affected Fingers or Toes by Dactylitis in Participants With Psoriatic Arthritis (PsA) at Weeks 12, 24, 36 and 52
Description: Each of the 10 fingers and 10 toes was evaluated for dactylitis. Score ranged from 0 to 20, where affected numbers of fingers and toes were evaluated.
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: finger or toes
Arm/Group | Etanercept
Number analyzed (Participants) | 254
finger or toes
  Week 12: number analyzed (Participants) | 65
  Week 12 | 1.4 (2.1)
  Week 24: number analyzed (Participants) | 58
  Week 24 | 0.7 (1.3)
  Week 36: number analyzed (Participants) | 52
  Week 36 | 0.7 (1.4)
  Week 52: number analyzed (Participants) | 49
  Week 52 | 0.6 (1.3)

38. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) in Participants With Plaque Psoriasis (PsO) at Weeks 12, 24, 36 and 52
Description: Combined assessment of lesion severity and area affected into single score. Body was divided into 4 sections: head, arms, trunk, legs. For each section, percent area of skin involved was estimated: 0= 0% involvement to 6= 90-100% involvement. Severity was estimated by clinical signs: erythema, induration, desquamation; scale: 0= none to 4= maximum. Final PASI = sum of severity parameters for each section*area score*weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4); total possible score range: 0= no disease to 72= maximal disease.
Time Frame: Baseline, Weeks 12, 24, 36, 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 70
units on a scale
  Baseline: number analyzed (Participants) | 66
  Baseline | 16.8 (10.1)
  Change at Week 12: number analyzed (Participants) | 64
  Change at Week 12 | -9.6 (10.3)
  Change at Week 24: number analyzed (Participants) | 55
  Change at Week 24 | -13.0 (10.6)
  Change at Week 36: number analyzed (Participants) | 43
  Change at Week 36 | -14.4 (10.9)
  Change at Week 52: number analyzed (Participants) | 40
  Change at Week 52 | -14.8 (11.0)

39. Secondary Outcome: Median Time to Achieve Psoriasis Area and Severity Index 75 (PASI 75) Response in Participants With Plaque Psoriasis (PsO)
Description: PASI: combined assessment of lesion severity & area affected into single score; range=0(no disease)-72(maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself & scores combined for final PASI. For each section % area of skin involved was estimated:0(0%) - 6(90-100%) & severity estimated by clinical signs of erythema, induration, desquamation; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor(head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4). PASI75: at least a 75 % reduction in PASI relative to Baseline.
Time Frame: Baseline up to Week 24
Population: as for outcome 5
Measure: Median (Standard Deviation); unit: days
Arm/Group | Etanercept
Number analyzed (Participants) | 70
days | 100 (85.6)

40. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Component Scores in Participants With Plaque Psoriasis (PsO)
Description: PASI: combined assessment of lesion severity & area affected into single score; range=0(no disease)-72(maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself & scores combined for final PASI. For each section % area of skin involved was estimated:0(0%) - 6(90-100%) & severity estimated by component score of erythema, induration, desquamation; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor(head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4).
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with PsO. "Number analyzed" signifies participants analyzed for this outcome measure at specified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 70
units on a scale
  Week 12, Erythema: number analyzed (Participants) | 63
  Week 12, Erythema | 1.4 (0.7)
  Week 12: Induration: number analyzed (Participants) | 63
  Week 12: Induration | 1.2 (0.7)
  Week 12: Desquamation: number analyzed (Participants) | 63
  Week 12: Desquamation | 1.1 (0.7)
  Week 24: Erythema: number analyzed (Participants) | 49
  Week 24: Erythema | 1.0 (0.7)
  Week 24: Induration: number analyzed (Participants) | 49
  Week 24: Induration | 0.9 (0.6)
  Week 24: Desquamation: number analyzed (Participants) | 49
  Week 24: Desquamation | 0.9 (0.7)
  Week 36: Erythema: number analyzed (Participants) | 41
  Week 36: Erythema | 0.7 (0.6)
  Week 36: Induration: number analyzed (Participants) | 41
  Week 36: Induration | 0.6 (0.5)
  Week 36: Desquamation: number analyzed (Participants) | 41
  Week 36: Desquamation | 0.6 (0.5)
  Week 52: Erythema: number analyzed (Participants) | 39
  Week 52: Erythema | 0.7 (0.7)
  Week 52: Induration: number analyzed (Participants) | 38
  Week 52: Induration | 0.5 (0.5)
  Week 52: Desquamation: number analyzed (Participants) | 39
  Week 52: Desquamation | 0.6 (0.6)

41. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Body Segment Scores in Participants With Plaque Psoriasis (PsO)
Description: PASI: combined assessment of lesion severity & area affected into single score; range=0(no disease)-72(maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself & scores combined for final PASI. For each section % area of skin involved was estimated:0(0%) - 6(90-100%) & severity estimated by clinical signs of erythema, induration, desquamation; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor(head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4).
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 70
units on a scale
  Week 12, Head: number analyzed (Participants) | 61
  Week 12, Head | 0.4 (0.8)
  Week 12: Trunk: number analyzed (Participants) | 62
  Week 12: Trunk | 1.6 (2.0)
  Week 12: Upper extremities: number analyzed (Participants) | 62
  Week 12: Upper extremities | 1.4 (1.6)
  Week 12: Lower extremities: number analyzed (Participants) | 62
  Week 12: Lower extremities | 3.5 (3.7)
  Week 24: Head: number analyzed (Participants) | 52
  Week 24: Head | 0.2 (0.5)
  Week 24: Trunk: number analyzed (Participants) | 51
  Week 24: Trunk | 0.6 (0.8)
  Week 24: Upper extremities: number analyzed (Participants) | 50
  Week 24: Upper extremities | 0.9 (1.0)
  Week 24: Lower extremities: number analyzed (Participants) | 52
  Week 24: Lower extremities | 2.3 (2.7)
  Week 36: Head: number analyzed (Participants) | 42
  Week 36: Head | 0.2 (0.4)
  Week 36: Trunk: number analyzed (Participants) | 42
  Week 36: Trunk | 0.5 (0.9)
  Week 36: Upper extremities: number analyzed (Participants) | 42
  Week 36: Upper extremities | 0.5 (0.5)
  Week 36: Lower extremities: number analyzed (Participants) | 42
  Week 36: Lower extremities | 1.5 (2.0)
  Week 52: Head: number analyzed (Participants) | 38
  Week 52: Head | 0.1 (0.3)
  Week 52: Trunk: number analyzed (Participants) | 39
  Week 52: Trunk | 0.5 (1.0)
  Week 52: Upper extremities: number analyzed (Participants) | 40
  Week 52: Upper extremities | 0.5 (0.5)
  Week 52: Lower extremities: number analyzed (Participants) | 39
  Week 52: Lower extremities | 1.4 (1.9)

42. Secondary Outcome: Dermatology Life Quality Index (DLQI) Total Score for Participants With Plaque Psoriasis (PsO) at Weeks 12, 24, 36 and 52
Description: The DLQI was a 10-item questionnaire that measures the impact of skin disease on participant's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The DLQI total score ranges from 0 (not at all) to 30 (very much): no effect at DLQI < 2; small effect at 2 <=DLQI <= 5; moderate effect at 6 <=DLQI <= 10; very large effect at 11<=DLQI <= 20; extremely large effect at 21 <= DLQI <= 30.
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 70
units on a scale
  Week 12: number analyzed (Participants) | 68
  Week 12 | 8.3 (7.4)
  Week 24: number analyzed (Participants) | 52
  Week 24 | 5.5 (5.8)
  Week 36: number analyzed (Participants) | 41
  Week 36 | 4.8 (5.5)
  Week 52: number analyzed (Participants) | 37
  Week 52 | 3.7 (4.6)

43. Secondary Outcome: Patient Assessment of Pruritus for Participants With Plaque Psoriasis (PsO) at Weeks 12, 24, 36 and 52
Description: Participant's assessment of pruritus measured on a 100 mm VAS ranging from 0 as "no Pruritus" to 100 as "most severe pruritus".
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 70
units on a scale
  Week 12: number analyzed (Participants) | 62
  Week 12 | 35.5 (30.9)
  Week 24: number analyzed (Participants) | 47
  Week 24 | 22.4 (23.8)
  Week 36: number analyzed (Participants) | 38
  Week 36 | 24.2 (26.6)
  Week 52: number analyzed (Participants) | 32
  Week 52 | 14.8 (15.8)

44. Other Pre Specified Outcome: Erythrocyte Sedimentation Rate (ESR) at Weeks 12, 24, 36 and 52
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm/hr. A higher rate is consistent with inflammation.
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. 'Number analyzed" signifies participants analyzed for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Etanercept
Number analyzed (Participants) | 1453
mm/hr
  Week 12: number analyzed (Participants) | 1139
  Week 12 | 19.7 (18.4)
  Week 24: number analyzed (Participants) | 938
  Week 24 | 19.4 (18.8)
  Week 36: number analyzed (Participants) | 800
  Week 36 | 18.4 (17.4)
  Week 52: number analyzed (Participants) | 741
  Week 52 | 18.2 (17.6)

45. Other Pre Specified Outcome: C-Reactive Protein (CRP) Levels at Weeks 12, 24, 36 and 52
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Etanercept
Number analyzed (Participants) | 1453
mg/L
  Week 12: number analyzed (Participants) | 1196
  Week 12 | 10.9 (33.9)
  Week 24: number analyzed (Participants) | 968
  Week 24 | 10.9 (37.4)
  Week 36: number analyzed (Participants) | 824
  Week 36 | 10.2 (31.4)
  Week 52: number analyzed (Participants) | 759
  Week 52 | 9.7 (30.3)

46. Other Pre Specified Outcome: Number of Participants With Rheumatoid Factor (RF) at Weeks 12, 24, 36 and 52
Description: RF is the auto antibody directed against immunoglobulin G (IgG) and its concentration is observed in human serum or plasma. RF value higher than 20 units per milliliter (U/mL) is considered positive.
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1383
Participants
  Week 12: number analyzed (Participants) | 1335
  Week 12 | 310
  Week 24: number analyzed (Participants) | 1114
  Week 24 | 259
  Week 36: number analyzed (Participants) | 958
  Week 36 | 208
  Week 52: number analyzed (Participants) | 866
  Week 52 | 173

47. Other Pre Specified Outcome: Anti-Cyclic Citrullinated Peptide (Anti-CCP) Antibodies at Weeks 12, 24, 36 and 52
Description: To assess the pharmacodynamics effect of etanercept on serum levels of autoantibodies, Anti-CCP antibodies levels were measured.
Time Frame: Weeks 12, 24, 36, 52
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with RA, AxS or PsA. "Number analyzed" signifies participants analyzed for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: unit per milliliter (U/mL)
Groups:
- Etanercept: All participants with RA, axSpA, or PsA taking etanercept in the routine treatment as per clinical practice and in line with summary of product characteristics clinical, were observed for a period of 12 months.
Arm/Group | Etanercept
Number analyzed (Participants) | 1383
unit per milliliter (U/mL)
  Week 12: number analyzed (Participants) | 94
  Week 12 | 236.2 (695.7)
  Week 24: number analyzed (Participants) | 77
  Week 24 | 202.2 (615.6)
  Week 36: number analyzed (Participants) | 68
  Week 36 | 178.6 (635.3)
  Week 52: number analyzed (Participants) | 52
  Week 52 | 176.2 (714.4)

48. Other Pre Specified Outcome: Number of Participants With Positive Human Leukocyte Antigen B27(HLA-B27) at Baseline for Participants With Axial Spondyloarthritis(axSpA)
Description: Participants with Axial Spondyloarthritis with Positive Human Leukocyte Antigen (HLA-B27) were reported.
Time Frame: Baseline
Population: PP set=all documented participants who were treated, had at least 1 post-baseline value, AE documented and no major protocol deviation. Overall number of participants analyzed signifies participants of PP set with axSpA.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 305
Participants | 223

49. Other Pre Specified Outcome: Number of Participants With Axial Spondyloarthritis (axSpA) Achieving Ankylosing Spondylitis Disease Activity Score (ASDAS) Less Than < 1.3 at Weeks 36 and 52
Description: as for outcome 6
Time Frame: Weeks 36, 52
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 305
Participants
  Week 36: number analyzed (Participants) | 131
  Week 36 | 35
  Week 52: number analyzed (Participants) | 137
  Week 52 | 32

50. Other Pre Specified Outcome: Number of Participants With Psoriatic Arthritis (PsA) Achieving Either 28 Joint Disease Activity Score (DAS28) Less Than < 2.6 or Meet Minimal Disease Activity (MDA) Criteria at Weeks 36 and 52
Description: as for outcome 7
Time Frame: Weeks 36, 52
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 254
Participants
  Week 36: number analyzed (Participants) | 181
  Week 36 | 93
  Week 52: number analyzed (Participants) | 161
  Week 52 | 87

51. Other Pre Specified Outcome: Number of Participants With Plaque Psoriasis (PsO) Achieving PASI75 Score or a PGA of "Clear" or "Almost Clear" And DLQI Total Score of 0 or 1 at Weeks 36 and 52
Description: as for outcome 5
Time Frame: Weeks 36, 52
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 70
Participants
  Week 36: number analyzed (Participants) | 48
  Week 36 | 13
  Week 52: number analyzed (Participants) | 44
  Week 52 | 14

52. Other Pre Specified Outcome: Number of Participants With Rheumatoid Arthritis (RA) Achieving 28 Joint Disease Activity Score (DAS28) Less Than (<) 2.6 at Weeks 36 and 52
Description: as for outcome 15
Time Frame: Weeks 36, 52
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 824
Participants
  Week 36: number analyzed (Participants) | 561
  Week 36 | 173
  Week 52: number analyzed (Participants) | 502
  Week 52 | 187

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: Same event may appear as both an AE & a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant & as non-serious in another participant, or one participant may have experienced both a serious & non-serious event during study. Treated set included all documented participants who were treated, had at least 1 post-baseline value & had an AE documented. All-cause mortality data included all anticipated & unanticipated deaths due to any cause.
Arm/Group | Etanercept
All-Cause Mortality (participants affected / at risk) | 5/1465
Serious Adverse Events (participants affected / at risk) | 151/1465
Other Adverse Events (participants affected / at risk) | 606/1465
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=1465)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Drug ineffective (General disorders) | 5
Condition aggravated (General disorders) | 16
Death (General disorders) | 3
Injection site reaction (General disorders) | 3
Pain (General disorders) | 2
Disease progression (General disorders) | 1
Disease recurrence (General disorders) | 1
Drug effect decreased (General disorders) | 1
Injection site erythema (General disorders) | 1
Injection site swelling (General disorders) | 1
Injection site warmth (General disorders) | 1
Implantation of medial unicondylar sliding prosthesis knee left (Surgical and medical procedures) | 1
Oedema peripheral (General disorders) | 1
Therapy non-responder (General disorders) | 1
Bronchitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 4
Diverticulitis (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Arthritis infective (Infections and infestations) | 1
Borrelia infection (Infections and infestations) | 1
Bronchitis bacterial (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Epididymitis (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Hepatitis e (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Mycobacterial infection (Infections and infestations) | 1
Nasal abscess (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Post procedural pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 2 — Only one participant died due to fall.
Femur fracture (Injury, poisoning and procedural complications) | 2
Meniscus injury (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Tracheal deviation (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Atrial fibrillation (Cardiac disorders) | 4
Arrhythmia (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 — Only one participant died due to pulmonary embolism.
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum haematoma (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 2
Crohn's disease (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral artery stenosis (Vascular disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 1
Vasculitis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Cholestasis (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatitis toxic (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Axonal neuropathy (Nervous system disorders) | 1
Facial paresis (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hepatic enzyme increased (Investigations) | 1
Renal function test abnormal (Investigations) | 1
Troponin increased (Investigations) | 1
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nephritis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Ureteric stenosis (Renal and urinary disorders) | 1
Inner ear disorder (Ear and labyrinth disorders) | 1
Vestibular disorder (Ear and labyrinth disorders) | 1
Drug hypersensitivity (Immune system disorders) | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2
Diplopia (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 1
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1
Goitre (Endocrine disorders) | 1
Restlessness (Psychiatric disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=1465)
Drug ineffective (General disorders) | 203
Condition aggravated (General disorders) | 35
Injection site erythema (General disorders) | 34
Injection site reaction (General disorders) | 22
Fatigue (General disorders) | 13
Injection site pruritus (General disorders) | 12
Pyrexia (General disorders) | 10
Drug effect decreased (General disorders) | 9
Pain (General disorders) | 8
Injection site hypersensitivity (General disorders) | 7
Oedema peripheral (General disorders) | 7
Injection site pain (General disorders) | 6
Injection site swelling (General disorders) | 6
Drug effect incomplete (General disorders) | 5
Injection site induration (General disorders) | 3
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 2
Chills (General disorders) | 2
Disease progression (General disorders) | 2
Injection site rash (General disorders) | 2
Local reaction (General disorders) | 2
Swelling (General disorders) | 2
Treatment failure (General disorders) | 2
Adverse event (General disorders) | 1
Asthenia (General disorders) | 1
Discomfort (General disorders) | 1
Disease recurrence (General disorders) | 1
Drug intolerance (General disorders) | 1
Face oedema (General disorders) | 1
Gait disturbance (General disorders) | 1
Hyperthermia (General disorders) | 1
Inflammation (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site discharge (General disorders) | 1
Injection site discolouration (General disorders) | 1
Injection site inflammation (General disorders) | 1
Injection site irritation (General disorders) | 1
Malaise (General disorders) | 1
Mucosal dryness (General disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Oedema (General disorders) | 1
Sensation of foreign body (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 62
Bronchitis (Infections and infestations) | 20
Respiratory tract infection (Infections and infestations) | 16
Upper respiratory tract infection (Infections and infestations) | 11
Infection (Infections and infestations) | 10
Herpes zoster (Infections and infestations) | 8
Sinusitis (Infections and infestations) | 8
Cystitis (Infections and infestations) | 7
Pulpitis dental (Infections and infestations) | 5
Tonsillitis (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 4
Gastrointestinal infection (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Conjunctivitis (Infections and infestations) | 2
Erysipelas (Infections and infestations) | 2
Fungal infection (Infections and infestations) | 2
Fungal skin infection (Infections and infestations) | 2
Paronychia (Infections and infestations) | 2
Rash pustular (Infections and infestations) | 2
Sinobronchitis (Infections and infestations) | 2
Skin candida (Infections and infestations) | 2
Subcutaneous abscess (Infections and infestations) | 2
Bacterial infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diabetic foot infection (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Groin abscess (Infections and infestations) | 1
Hepatitis e (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Papilloma viral infection (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Superinfection bacterial (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Urinary tract infection enterococcal (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 16
Erythema (Skin and subcutaneous tissue disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 12
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 5
Psoriasis (Skin and subcutaneous tissue disorders) | 5
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 4
Skin disorder (Skin and subcutaneous tissue disorders) | 4
Skin reaction (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 4
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 3
Skin irritation (Skin and subcutaneous tissue disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Vascular skin disorder (Skin and subcutaneous tissue disorders) | 1
Xanthelasma (Skin and subcutaneous tissue disorders) | 1
Infected bite (Infections and infestations) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Joint swelling (Musculoskeletal and connective tissue disorders) | 5
Bursitis (Musculoskeletal and connective tissue disorders) | 4
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4
Joint effusion (Musculoskeletal and connective tissue disorders) | 3
Limb discomfort (Musculoskeletal and connective tissue disorders) | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3
Synovitis (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Enthesopathy (Musculoskeletal and connective tissue disorders) | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2
Osteitis (Musculoskeletal and connective tissue disorders) | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2
Tendon disorder (Musculoskeletal and connective tissue disorders) | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Dactylitis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1
Mastication disorder (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 12
Abdominal discomfort (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Loose tooth (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Steatorrhoea (Gastrointestinal disorders) | 1
Tongue discomfort (Gastrointestinal disorders) | 1
Tooth disorder (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 4
Carpal tunnel syndrome (Nervous system disorders) | 3
Burning sensation (Nervous system disorders) | 2
Head discomfort (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Balance disorder (Nervous system disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 1
Complex regional pain syndrome (Nervous system disorders) | 1
Coordination abnormal (Nervous system disorders) | 1
Cubital tunnel syndrome (Nervous system disorders) | 1
Intercostal neuralgia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Movement disorder (Nervous system disorders) | 1
Spinal cord disorder (Nervous system disorders) | 1
Trigeminal neuralgia (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 1
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 5
Ligament sprain (Injury, poisoning and procedural complications) | 3
Wound (Injury, poisoning and procedural complications) | 3
Contusion (Injury, poisoning and procedural complications) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Inflammation of wound (Injury, poisoning and procedural complications) | 1
Ligament injury (Injury, poisoning and procedural complications) | 1
Maternal exposure before pregnancy (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Liver function test increased (Investigations) | 2
Transaminases increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Blood thyroid stimulating hormone abnormal (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Heart rate increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Intraocular pressure increased (Investigations) | 1
Renal function test abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
Depression (Psychiatric disorders) | 8
Sleep disorder (Psychiatric disorders) | 2
Aggression (Psychiatric disorders) | 1
Apathy (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Somatic symptom disorder (Psychiatric disorders) | 1
Iritis (Eye disorders) | 4
Visual impairment (Eye disorders) | 2
Eye swelling (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Vitamin d deficiency (Metabolism and nutrition disorders) | 4
Gout (Metabolism and nutrition disorders) | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Metabolic syndrome (Metabolism and nutrition disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Increased tendency to bruise (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 2
Granulocytopenia (Blood and lymphatic system disorders) | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Bladder disorder (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Leukocyturia (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 2
Extrasystoles (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Hypersensitivity (Immune system disorders) | 5
Anaphylactic reaction (Immune system disorders) | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Deafness (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1
Uterine haematoma (Reproductive system and breast disorders) | 1
Peripheral venous disease (Vascular disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT02486302/Prot_SAP_000.pdf